CLINICAL TRIAL: NCT07112235
Title: Using Multiomics to Define Mechanisms of RhinoVirus-induced Chronic Obstructive Pulmonary Disease Exacerbations to Develop Novel Therapies and Therapeutic Targets
Acronym: MRVCOPD
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 172255; MR/Z504531/1 (Other Grant/Funding Number: UKRI Medical Research Council)
Record Dates: First submitted 2025-07-11; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Rhinovirus Infection; Exacerbation of COPD
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Exacerbation; Multiomics; Rhinovirus; Viral challenge study
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD Subjects: Participants who meet the diagnostic criteria for COPD
  Interventions: Biological: Rhinovirus-A16
- Non-Smoking Controls: Participants who do not meet COPD diagnostic criteria, and who do not have a significant smoking history
  Interventions: Biological: Rhinovirus-A16
- Smoking Controls: Participants who do not meet COPD diagnostic criteria, and who do have a significant smoking history
  Interventions: Biological: Rhinovirus-A16

INTERVENTIONS:
Biological: Rhinovirus-A16 — Nasal inoculation with a dose equivalent to 100 TCID50 of rhinovirus-A16 inoculum will be administered to all participants in the study

SUMMARY:
The goal of this study is to examine exacerbations of chronic obstructive pulmonary disease (COPD) caused by a common cold virus called rhinovirus, to identify new treatments. Exacerbations are flare-ups of respiratory symptoms which are a major cause of ill health in people with COPD, and are most commonly caused by viruses.

The main questions the study aims to answer are:

* What processes in the body occur in response to rhinovirus infection, and do the differences between people with COPD and healthy volunteers explain why people with COPD develop more severe illness and exacerbations?
* Can treatments be identified that target these processes to reduce the severity and frequency of exacerbations in people with COPD?

The study will compare eligible participants with COPD to healthy volunteers, and will involve intentionally infecting each participant with rhinovirus in a controlled environment. They will undergo baseline investigations prior to infection including a first bronchoscopy. Post-infection each participant will undergo a range of tests, including a second bronchoscopy, to compare how processes in the body, and especially the lungs, differ between people who do and do not have COPD.

DETAILED DESCRIPTION:
Study Rationale:

The investigators aim to understand the biological mechanisms that underlie exacerbations of Chronic Obstructive Pulmonary Disease (COPD) to drive the discovery of new treatments.

COPD is the 4th leading cause of death worldwide, causing 3.5 million deaths in 2021. Acute exacerbations of COPD (AECOPD) involve sudden flare-ups of symptoms, commonly triggered by viral infections, and are the major cause of COPD morbidity, mortality and healthcare costs. Developing new treatments for AECOPD requires a better understanding of the processes occurring in the lungs, before and during exacerbations. Naturally-occurring AECOPD are challenging to study in a way that allows reliable measurement of disease mechanisms, and repeated lung sampling can be impractical and potentially dangerous.

The investigators have therefore developed a human rhinovirus challenge experimental model of AECOPD. This involves infecting participants with a common cold virus called rhinovirus (RV). These studies have demonstrated that RV causes mild-to-moderate exacerbations in 95% of COPD subjects, that confounding factors can be controlled to take reliable measurements, and that repeated sampling of the lungs and respiratory tract can safely and easily be performed in a controlled research environment.

The investigators will compare people who have COPD with people who do not have COPD, including smokers and non-smokers, to identify the processes important in COPD. Researchers will measure a range of clinical and scientific outcomes, using cutting-edge 'multiomics' techniques to understand mechanisms in RV-induced AECOPD to an extent that has not been achieved before.

The crucial information that this study generates will be used to identify new treatments to reduce the frequency and severity of AECOPD. Data will be made publicly available for others to use and analyse, and will be integrated with other databases to maximise the scientific benefit that is gained from our participants' contribution to the project.

End of Study:

Follow up period of 42 days

Study Centres:

There will be 1 study centre: Imperial College Healthcare NHS Trust

Study Intervention:

All participants will be inoculated intra-nasally with rhinovirus-A16

Study Sample Size:

25 participants with mild/moderate COPD, 13 smoking controls, 12 non-smoking controls.

Study procedures

* Screening visit: lung function tests (FEV1, FVC and PEF), height and weight/BMI, Medical and surgical history, drug history, pregnancy test for females with childbearing potential, blood sample.
* Baseline visit: Baseline questionnaires, initiation of daily diary card, blood tests (including for haematology, biochemistry and coagulation), vital signs, physical examination, nasosorption, nasal lavage, nasal and oropharyngeal swabs, sputum collection, chest x-ray, electrocardiogram, lung function tests (FEV1, FVC, PEF), FeNO, airway oscillometry and skin prick testing.
* Baseline bronchoscopy: Bronchoscopy including bronchosorption, bronchioalveolar lavage, bronchial brushings and bronchial biopsies.
* Visit Day 0: Viral inoculation visit: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection, urine collection and intranasal RV-A16 challenge
* Visit Day 1: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection, urine collection
* Visit Day 2: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), nasosorption, nasal and oropharyngeal swabs, nasal lavage, urine collection.
* Visit Day 3: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection, urine collection
* Visit Day 4: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), nasosorption, nasal and oropharyngeal swabs, nasal lavage, urine collection.
* Visit Day 5: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection, urine collection
* Visit Day 7 and Bronchoscopy: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, urine collection and bronchoscopy including bronchosorption, bronchioalveolar lavage, bronchial brushings and bronchial biopsies
* Visit Day 9: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection, urine collection.
* Visit Day 12: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection, urine collection.
* Visit Day 15: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection, urine collection.
* Visit Day 21: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection.
* Visit Day 42: Vital signs, physical examination, lung function tests (FEV1, FVC, PEF), airway oscillometry, FeNO, nasosorption, nasal and oropharyngeal swabs, nasal lavage, blood sampling, sputum collection. On completion of this visit the participant will have finished the study and will no longer be enrolled.

ELIGIBILITY:
Inclusion Criteria for COPD subjects

* Male or female sex
* Age ≥40 years and ≤75 years at the time of signing the consent form
* Medical history or clinical diagnosis of COPD
* Significant smoking history, defined as:

  * Cumulative smoking history of at least 20 pack years
  * Permitted to currently use, or have history of use of, e-cigarettes/vapes
* COPD spirometry criteria:

  * Post bronchodilator FEV1 of <80% and ≥50% predicted for age and height (equivalent to GOLD criteria stage 2 for 'Moderate' severity COPD9)
  * Post-bronchodilator FEV1/FVC ratio <0.7
  * β-agonist reversibility: an improvement of less than 12% predicted FEV1 and less than 200mL after 200 micrograms of salbutamol or equivalent short acting beta-2 agonist bronchodilator.
* History of acute exacerbations of COPD as defined by the participant answering "yes" to the question: "do your COPD symptoms get noticeably worse when you catch a cold?"
* Clinically stable with no COPD exacerbations within 8 weeks prior to enrolment
* Permitted to take short and long-acting bronchodilators including beta agonists and muscarinic antagonist inhalers
* Co-morbidity criteria:

  * Permitted to have a past medical history of asthma, allergic rhinitis and seasonal rhinitis, but not currently active within 8 weeks prior to enrolment
  * Absence of current or previous history of significant respiratory disease, other than COPD, asthma and allergic rhinitis
* Permitted to have a positive skin test for atopy

Inclusion Criteria for non-smoking controls

* Male or female sex
* Age ≥ 40 years and ≤ 75 years at the time of signing the consent form
* No history or clinical diagnosis of COPD
* No significant smoking history, defined as:

  * Less than 5 pack year cumulative smoking history
  * Has not smoked or used e-cigarettes/vapes in the last 1 year
* Controls spirometry criteria

  * FEV1 of ≥80% predicted for age and height
  * FEV1/FVC ratio ≥0.7
* Co-morbidity criteria:

  * Permitted to have a past medical history of asthma, allergic rhinitis and seasonal rhinitis, but not currently active in the 8 weeks prior to enrolment
  * Absence of current or previous history of significant respiratory disease, other than asthma and allergic rhinitis
* Permitted to have a positive skin test for atopy.

Inclusion Criteria for smoking controls

• Identical to non-smoking controls, with the exception of smoking history:

* Cumulative smoking history of at least 20 pack years.
* Permitted to currently use, or have history of use of, e-cigarettes/vapes

Exclusion Criteria:

* Participants with other causes of chronic airflow limitation, including but not limited to:

  * Bronchiectasis including cystic fibrosis
  * Bronchiolitis obliterans
  * Carcinoma of the bronchus
  * Fibrosis such as tuberculosis (TB), idiopathic pulmonary fibrosis
* Presence of any significant systemic disease, that in the opinion of the investigator would (a) make participation in the study unduly risky, or (b) significantly interfere with important outcomes being measured.

  * For example, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric conditions.
* Pregnant, planning to become pregnant, testing positive for pregnancy at the screening visit test, or nursing females during and within 30 days of treatment.
* Treatment with oral, inhaled or nasal corticosteroids within 8 weeks prior to enrolment.
* Treatment with antibiotics in the 8 weeks preceding enrolment.
* Treatment with nasal medications, anti-leukotrienes, anti-histamine at the time of the study.
* Presence (at screening) of serum rhinovirus-A16 neutralising antibodies in a titre >1:2.
* Individuals with close contact to at risk patient group, including:

  * Infants (less than 6 months);
  * The extremely elderly or infirm;
  * Pregnant and/or breastfeeding women;
  * Patients with immunosuppression (e.g., human immunodeficiency virus (HIV), transplant recipients on anti-rejection medications, those undergoing chemo- or immuno-therapy).
  * Other factors that in the opinion of the investigator are considered a risk.
* Participation in other clinical research studies that, in the opinion of the investigator, would (a) make participation in the study unduly risky, or (b) significantly interfere with important outcomes being measured in this or other studies, or (c) present an unacceptable visit burden to the participant.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit participants that respond to advertisement or invitations to participate in the study, that meet the eligibility criteria, and whom are willing and able to consent to take part in this study which involves 15 study visits over the course of 7-10 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Lower Respiratory Symptom Score (LRSS) | Participants will record this score daily, from the date of the baseline visit to the final day of their involvement in the study (expected to be day 42).
  Participants will be asked to record their lower respiratory tract symptom scores daily prior to and in the 42 days following viral infection with rhinovirus A-16. Participants will rate their shortness of breath, wheeze, cough, sputum quality and quantity. Total score ranges from 0-17, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Upper Respiratory Symptom Score (URSS) | Participants will record this score daily, from the date of the baseline visit to the final day of their involvement in the study (expected to be day 42).
  Participants will be asked to record their upper respiratory tract symptom scores daily prior to and in the 42 days following viral infection with rhinovirus A-16. Participants will rate their symptoms of cough, sneezing, runny nose, blocked nose, headache, sore throat, malaise, and fever. Total score ranges from 0-24, with higher scores indicating more severe symptoms.
EXAcerbations of Chronic pulmonary disease Tool-Patient Reported Outcomes (EXACT-PRO) | Participants will record this score daily, from the date of the baseline visit to the final day of their involvement in the study (expected to be day 42).
  Participants will be asked to record scores for symptoms commonly experienced in COPD exacerbations daily prior to and in the 42 days following viral infection with rhinovirus A-16. Participants will rate their chest congestion, cough, mucus quality and quantity, chest discomfort, chest tightness, general breathlessness, shortness of breath whilst performing personal care, indoor activities and outside errands, tiredness, sleep, and anxiety. Total score ranges from 0-100, with higher scores indicating more severe symptoms.
Forced Expiratory Volume in 1 second (FEV1) | FEV1 will be measured at baseline, on day 0 and every following visit (days 1, 2, 3, 4, 5, 7, 9, 12, 15, 21 and 42).
  Investigators will perform lung function/spirometry at baseline, immediately prior to inoculation, and at every clinical visit after RV inoculation. The primary measure of lung function will be the forced expiratory volume in 1 second (FEV1), which is a measure of larger airway patency and is impaired in COPD and further impaired in exacerbations of COPD.
Airway Oscillometry | Investigators will measure participants' airway oscillometry at baseline and clinical visits days 0, 3, 5, 9, 12, 15, 21, 42.
  Airway oscillometry is a technique used to measure airflow and patency of the airways, and is a more sensitive measure of small airway dysfunction than spirometry and FEV1.
Fractional exhaled nitric oxide (FeNO) | Investigators will measure participants' FeNO at baseline and at clinical visits on days 0, 3, 5, 9, 12, 15, 21, 42
  FeNO measures the concentration of nitric oxide in exhaled breath from subjects, which is an indicator of airway inflammation.
Viral load | Nasal lavage and nasal swabs will be performed at baseline and on all post inoculation visits. Sputum will be collected at baseline and on visits on days 0, 1, 3, 5, 9, 12, 15, 21 and 42. BAL will be acquired via bronchoscopy at baseline and day 7.
  Investigator will measure the load of rhinovirus-A16 via quantitative PCR in nasal lavage, nasal swabs, sputum and bronchoalveolar lavage (BAL) acquired from participants.
Cellular interferon response to rhinovirus infection | Studies performed on cells extracted at baseline (pre-inoculation) bronchoscopy.
  Investigators will perform laboratory quantification of immune and epithelial cell interferon response to rhinovirus response in vivo.
Immunological response to rhinovirus infection | Blood will be taken at baseline and at visits on day 0, 1, 3, 5, 7, 9, 12, 15, 21, 42. Nasosorption will be performed at baseline and all visits post inoculation. Bronchial biopsies, bronchosorption will be via bronchoscopy at baseline and day 7.
  Investigators will measure the number of inflammatory cells in bronchial epithelium and in peripheral blood (via flow cytometry of peripheral blood, and single cell RNA sequencing and spatial transcriptomics of bronchial biopsies), and in the expression of alarmins and cytokines on nasal and bronchial epithelium (via proteomic analysis of naso- and broncho-sorption samples).
Evaluation of the respiratory microbiome | Sputum will be collected at baseline and on visits on days 0, 1, 3, 5, 9, 12, 15, 21 and 42. BAL will be acquired via bronchoscopy at baseline and day 7.
  Microbial culture and detailed microbiome assessment of sputum samples and bronchoalveolar lavage samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian L Johnston, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We may share results from this study with anonymised databases, for example the Human Lung Cell Atlas, whereby the valuable data that our participants have generously provided can lead to the maximum scientific gain. However if this does proceed, then the data will be carefully anonymised and reviewed to ensure that it does not contain personally identifiable data, so that our participants retain the strictest confidentiality and privacy.